CLINICAL TRIAL: NCT01311687
Title: A Phase 3, Muticenter, Randomized, Open-label Study to Compare the Efficacy and Safety of Pomalidomide in Combination With Low-dose Dexamethasone Versus High-dose Dexamethasone in Subjects With Refractory or Relapsed and Refractory Multiple Myeloma
Brief Title: A Phase 3, Multicenter, Randomized, Open-Label Study to Compare the Efficacy and Safety of Pomalidomide in Combination With Low-Dose Dexamethasone Versus High-Dose Dexamethasone in Subjects With Refractory Multiple Myeloma or Relapsed and Refractory Multiple Myeloma and Companion Study
Acronym: NIMBUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-MM-003; 2010-019820-30 (EudraCT Number)
Record Dates: First submitted 2011-03-08; First posted 2011-03-09 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-09

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; Relapsed Multiple Myeloma; Relapsed and Refractory Multiple Myeloma; Refractory Myeloma; Resistant Multiple Myeloma; Treatment-resistant Multiple Myeloma; Pomalidomide; Lenalidomide-resistant; Bortezomib-resistant
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Recurrence | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pomalidomide + Low-Dose Dexamethasone (Experimental): Participants received 4 mg pomalidomide administered by mouth on Days 1 to 21 of each 28-day treatment cycle and 40 mg dexamethasone (or 20 mg for participants > 75 years of age) administered by mouth once per day on Days 1, 8, 15, and 22 of each 28-day cycle until disease progression.
  Interventions: Drug: pomalidomide; Drug: Dexamethasone
- High-Dose Dexamethasone (Active Comparator): Participants received 40 mg dexamethasone (or 20 mg for participants > 75 years of age) administered by mouth once per day on Days 1 to 4, 9 to 12, and 17 to 20 of each 28-day treatment cycle until disease progression.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: pomalidomide — 4 mg pomalidomide capsules administered orally
  Other Names: CC-4047; Pomalyst®
  Arms: Pomalidomide + Low-Dose Dexamethasone
Drug: Dexamethasone — 40 mg dexamethasone (or 20 mg for participants > 75 years of age) tablets administered orally

SUMMARY:
The purpose of this study is to compare efficacy and safety of pomalidomide in combination with low-dose dexamethasone versus high-dose dexamethasone in subjects with refractory or relapsed and refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥ 18 years of age
* Subjects must have documented diagnosis of multiple myeloma and have measurable disease
* Subjects must have undergone prior treatment with ≥ 2 treatment lines of anti-myeloma therapy
* Subjects must have either refractory or relapsed and refractory disease defined as documented disease progression during or within 60 days of completing their last myeloma therapy
* All subjects must have received at least 2 consecutive cycles of prior treatment that included lenalidomide and bortezomib
* All subjects must have failed treatment with both lenalidomide and bortezomib in one of the following ways: 1) Documented progressive disease on or within 60 days of completing treatment with lenalidomide and/or bortezomib, or 2) In case of prior response [≥ partial response (PR)] to lenalidomide or bortezomib, subjects must have relapsed within 6 months after stopping treatment with lenalidomide and/or bortezomib-containing regimens, or 3) Subjects who have not had a ≥ minimal response (MR) and have developed intolerance/toxicity after a minimum of two cycles of lenalidomide- and/or bortezomib-containing regimen
* Patients must have received adequate prior alkylator therapy
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Females of childbearing potential (FCBP) must not become pregnant for 28 days prior to initiation of study drug, during the study, and for 28 days after discontinuation
* Females must agree to abstain from breastfeeding during study participation and 28 days after study drug discontinuation
* Males must agree to use a latex condom during any sexual during the study and for 28 days following discontinuation from this study
* Males must also agree to refrain from donating semen or sperm while on pomalidomide and for 28 days after discontinuation from this study

Exclusion Criteria:

* Any of the following laboratory abnormalities:

  * Absolute neutrophil count (ANC) < 1,000/μL
  * Platelet count < 75,000/ μL for subjects in whom < 50% of bone marrow nucleated cells are plasma cells
  * Creatinine clearance < 45 mL/min
  * Corrected serum calcium > 14 mg/dL
  * Hemoglobin ≤ 8 g/dL
  * Serum glutamic oxaloacetic transaminase (SGOT)/ aspartate aminotransferase (AST) or transaminase, serum glutamic pyruvic (SGPT)/ alanine aminotransferase (ALT) > 3.0 x upper limit of normal (ULN)
  * Serum total bilirubin > 2.0 mg/dL
* Previous therapy with pomalidomide
* Hypersensitivity to thalidomide, lenalidomide, or dexamethasone
* Resistance to high-dose dexamethasone used in the last line of therapy
* Peripheral neuropathy ≥ Grade 2
* Subjects who received an allogeneic bone marrow or allogeneic peripheral blood stem cell transplant
* Subjects who are planning for or who are eligible for stem cell transplant
* Subjects with any one of the following: 1) Congestive heart failure, 2) Myocardial infarction within 12 months prior to starting study treatment, 3) Unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris
* Subjects who received any of the following within the last 14 days of initiation of study treatment: 1) Plasmapheresis, 2) Major surgery, 3) Radiation therapy, 4) Use of any anti-myeloma drug therapy
* Use of any investigational agents within 28 days or 5 half-lives (whichever is longer) of treatment
* Subjects with conditions requiring chronic steroid or immunosuppressive treatment
* Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
* Incidence of gastrointestinal disease that may significantly alter the absorption of pomalidomide
* Subjects unable or unwilling to undergo antithrombotic prophylactic treatment
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subjects from signing the informed consent form
* Pregnant or breastfeeding females
* Known human immunodeficiency virus (HIV) positivity or active infectious hepatitis A, B, or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2011-03-11 (Actual); Primary Completion 2013-03-01 (Actual); Study Completion 2017-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Sternas, MD, PhD, Study Director — Celgene
Locations (94):
- Mayo Clinic, Rochester, Minnesota, United States
- Australia (10):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Institute, East Melbourne, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Princess Alexandra Hospital, Brisbane
  - Royal Prince Alfred Hospital, Camperdown
  - Alfred hospital, Melbourne
  - Sir Charles Gairdner Hospital, Nedlands
  - Calvary Mater Hospital, Waratah
  - Border Medical Oncology, Wodonga
  - Wollongong Hospital, Wollongong
- Belgium (3):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHU UCL Mont-Godinne-Dinant asbl, Yvoir
- Canada (10):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - James Cancer Hospital, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - University Health Network, Toronto, Ontario
  - Maisonneuve Rosemont, Montreal, Quebec
  - Royal Victoria Hospital McGill Department of Oncology(RVH), Montreal, Quebec
  - Sir Mortimer B. Davis - Jewish Genl, Montreal, Quebec
- Charles University General Hospital, Prague, Czechia
- Denmark (4):
  - Hæmatologisk afd. B Aalborg Sygehus Syd, Aalborg
  - Aarhus University Hospital, Arhus C
  - Odense Universitetshospital, Odense C
  - Vejle Hospital, Vejle
- France (13):
  - CHU d'Angers, Angers
  - Centre Hospitalier de la cote basque, Bayonne
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - CHRU de Lille FR, Lille
  - Institut Paoli-Calmettes, Marseille
  - CHRU Nantes, Nantes
  - Hopital Saint-Louis, Paris
  - CHU Hôpital St-Antoine, Paris
  - CHRU - Hopital du Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Bretonneau, Tours
  - Hopital Purpan, Tulouse Cedex 9
  - CHU Nancy, Vandœuvre-lès-Nancy
- Germany (9):
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Universitatsklinikum Essen, Essen
  - Askepios Klinik St. Georg, Hamburg
  - Universitatsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Jena, Jena
  - Universitatsklinikum Leipzig, Leipzig
  - University of Tubingen, Tübingen
  - Universitatsklinikum Ulm, Ulm
  - Universitatsklinikum Wurzburg, Würzburg
- Alexandra General Hospital of Athens, Athens, Greece
- Italy (9):
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Clinica Ematologica- A.O.U. San Martino, Genova
  - Oncoematologia, Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - AOU San Luigi Gonzaga, Orbassano
  - Universita degli Studi di Padova, Padua
  - Hospital Clinic, Placenza
  - Servizio di Ematologia, A.O. - Arcispedale S.Maria Nuova, Reggio Emilia
  - Univerita La Sapienza Dipartimento di Biotecnologie Cellulari ed Ematologia, Rome
  - Azienda Ospedaliera San Giovanni Battista, Torino
- Netherlands (3):
  - VU University Medical Center, Amsterdam
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Russia (4):
  - State Institution Hematological Research, Centre of Russian Academy of Medical Science, Moscow
  - State Institution Moscow Regional Research Clinical Institute, Moscow
  - St. Petersburg Research Institute of Hematology and Blood Transfusion, Saint Petersburg
  - State Educational Institution, Saint Petersburg State Medical University, Saint Petersburg
- Spain (8):
  - Hospital Universitari Germans Trias i Pujol, Badalona (Barcelona)
  - Hospital Clinic Provincial de Barcelona, Barcelona
  - Hospital de La Princesa, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Donostia, San Sebastián (Guipuzcoa)
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital de la Fe, Valencia
- Sweden (5):
  - Department of Hematology Hematology Centre, Gothenburg
  - University Hospital in Lund, Lund
  - Karolinska University Hospital Huddinge, Stockholm
  - Karolinska University Hospital, Stockholm
  - Overlakare Medocomcentrum, hematologi, Uppsala
- Switzerland (3):
  - Medizinische Universitatsklinik, Bern
  - Hopitaux Universitaires de Geneve-HUG, Geneva
  - UniversitatSspital Zurich, Zurich
- United Kingdom (10):
  - Royal Bournemouth Hospital, Bournemouth
  - St James's University Hospital, Leeds
  - St.Bartholomew's Hospital, London
  - King's College Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Derriford Hospital, Plymouth
  - Royal Hallamshire HospitalSheffield Teaching Hospitals NHS Trust, Sheffield
  - The Royal Marsden Hospital, Sutton-Surrey
  - The Royal Wolverhampton Hospital NHS Trust, Wolverhampton

REFERENCES:
- [Result] Moreau P, Weisel KC, Song KW, Gibson CJ, Saunders O, Sternas LA, Hong K, Zaki MH, Dimopoulos MA. Relationship of response and survival in patients with relapsed and refractory multiple myeloma treated with pomalidomide plus low-dose dexamethasone in the MM-003 trial randomized phase III trial (NIMBUS). Leuk Lymphoma. 2016 Dec;57(12):2839-2847. doi: 10.1080/10428194.2016.1180685. Epub 2016 May 13. PMID 27173785
- [Result] Miguel JS, Weisel K, Moreau P, Lacy M, Song K, Delforge M, Karlin L, Goldschmidt H, Banos A, Oriol A, Alegre A, Chen C, Cavo M, Garderet L, Ivanova V, Martinez-Lopez J, Belch A, Palumbo A, Schey S, Sonneveld P, Yu X, Sternas L, Jacques C, Zaki M, Dimopoulos M. Pomalidomide plus low-dose dexamethasone versus high-dose dexamethasone alone for patients with relapsed and refractory multiple myeloma (MM-003): a randomised, open-label, phase 3 trial. Lancet Oncol. 2013 Oct;14(11):1055-1066. doi: 10.1016/S1470-2045(13)70380-2. Epub 2013 Sep 3. PMID 24007748
- [Derived] Siegel DS, Weisel KC, Dimopoulos MA, Baz R, Richardson P, Delforge M, Song KW, San Miguel JF, Moreau P, Goldschmidt H, Cavo M, Jagannath S, Yu X, Hong K, Sternas L, Zaki M, Palumbo A. Pomalidomide plus low-dose dexamethasone in patients with relapsed/refractory multiple myeloma and moderate renal impairment: a pooled analysis of three clinical trials. Leuk Lymphoma. 2016 Dec;57(12):2833-2838. doi: 10.1080/10428194.2016.1177181. Epub 2016 Jun 7. PMID 27267105
- [Derived] Weisel KC, Dimopoulos MA, Moreau P, Lacy MQ, Song KW, Delforge M, Karlin L, Goldschmidt H, Banos A, Oriol A, Alegre A, Chen C, Cavo M, Garderet L, Ivanova V, Martinez-Lopez J, Knop S, Yu X, Hong K, Sternas L, Jacques C, Zaki MH, San Miguel J. Analysis of renal impairment in MM-003, a phase III study of pomalidomide + low - dose dexamethasone versus high - dose dexamethasone in refractory or relapsed and refractory multiple myeloma. Haematologica. 2016 Jul;101(7):872-8. doi: 10.3324/haematol.2015.137083. Epub 2016 Apr 14. PMID 27081177
- [Derived] Dimopoulos MA, Weisel KC, Song KW, Delforge M, Karlin L, Goldschmidt H, Moreau P, Banos A, Oriol A, Garderet L, Cavo M, Ivanova V, Alegre A, Martinez-Lopez J, Chen C, Spencer A, Knop S, Bahlis NJ, Renner C, Yu X, Hong K, Sternas L, Jacques C, Zaki MH, San Miguel JF. Cytogenetics and long-term survival of patients with refractory or relapsed and refractory multiple myeloma treated with pomalidomide and low-dose dexamethasone. Haematologica. 2015 Oct;100(10):1327-33. doi: 10.3324/haematol.2014.117077. Epub 2015 Aug 6. PMID 26250580
- [Derived] San Miguel JF, Weisel KC, Song KW, Delforge M, Karlin L, Goldschmidt H, Moreau P, Banos A, Oriol A, Garderet L, Cavo M, Ivanova V, Alegre A, Martinez-Lopez J, Chen C, Renner C, Bahlis NJ, Yu X, Teasdale T, Sternas L, Jacques C, Zaki MH, Dimopoulos MA. Impact of prior treatment and depth of response on survival in MM-003, a randomized phase 3 study comparing pomalidomide plus low-dose dexamethasone versus high-dose dexamethasone in relapsed/refractory multiple myeloma. Haematologica. 2015 Oct;100(10):1334-9. doi: 10.3324/haematol.2015.125864. Epub 2015 Jul 9. PMID 26160879
- [Derived] Weisel K, Dimopoulos M, Song KW, Moreau P, Palumbo A, Belch A, Schey S, Sonneveld P, Sternas L, Yu X, Amatya R, Gibson CJ, Zaki M, Jacques C, San Miguel J. Pomalidomide and Low-Dose Dexamethasone Improves Health-Related Quality of Life and Prolongs Time to Worsening in Relapsed/Refractory Patients With Multiple Myeloma Enrolled in the MM-003 Randomized Phase III Trial. Clin Lymphoma Myeloma Leuk. 2015 Sep;15(9):519-30. doi: 10.1016/j.clml.2015.05.007. Epub 2015 Jun 6. PMID 26149712
- [Derived] Song KW, Dimopoulos MA, Weisel KC, Moreau P, Palumbo A, Belch A, Schey S, Sonneveld P, Sternas L, Yu X, Amatya R, Monzini MS, Zaki M, Jacques C, San Miguel J. Health-related quality of life from the MM-003 trial of pomalidomide plus low-dose dexamethasone versus high-dose dexamethasone in relapsed and/or refractory multiple myeloma. Haematologica. 2015 Feb;100(2):e63-7. doi: 10.3324/haematol.2014.112557. Epub 2014 Nov 25. No abstract available. PMID 25425684

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 93 sites: 68 sites in Europe, 10 sites in Australia, 10 sites in Canada, 4 sites in Russia, and 1 site in the United States (US) from 18 March 2011 to 29 August 2017.
Pre-assignment Details: Participants were randomized in a 2:1 ratio. Treatment phase discontinuation occurred when a participant had confirmed progressive disease. Participants who did not progress but who were intolerant to treatment, or no longer wished to receive study treatment entered the progression-free survival (PFS) follow-up period until disease progression.
Groups:
- Pomalidomide Plus Low-Dose Dexamethasone: Participants received 4 mg pomalidomide administered by mouth on Days 1-21 of each 28-day treatment cycle and 40 mg dexamethasone (participants > 75 years of age received 20 mg dexamethasone) administered by mouth once per day on Days 1, 8, 15, and 22 of a 28-day cycle until disease progression.
- High-Dose Dexamethasone (HD-Dex): Participants received 40 mg dexamethasone (participants > 75 years of age received 20 mg dexamethasone) administered by mouth once per day on Days 1 through 4, 9 through 12, and 17 through 20 of a 28-day cycle until disease progression.
Period: Treatment Phase
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone (HD-Dex)
Started | 302 | 153
Received Study Drug | 300 | 150
Crossed-over to Pomalidomide | 0 (Not applicable to participants initially randomized to receive pomalidomide) | 11 (After Amendment 4 participants still on HD-Dex treatment were permitted to crossover to pomalidomide)
Completed (Completed represents participants who discontinued from study treatment) | 302 | 153
Not Completed | 0 | 0
Period: PFS Follow-up Phase
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone (HD-Dex)
Started | 11 | 8
Crossed-over to Pomalidomide (After Amendment 4 participants still on HD-Dex treatment were permitted to crossover to pomalidomide) | 11 | 0
Completed (Completed represents participants who discontinued from PFS follow-up) | 11 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population (all participants who were randomized, regardless of whether they received study treatment or not)
Groups:
- High-Dose Dexamethasone: Participants received 40 mg dexamethasone (participants > 75 years of age received 20 mg dexamethasone) administered by mouth once per day on Days 1 through 4, 9 through 12, and 17 through 20 of a 28-day cycle until disease progression.
- Total: Total of all reporting groups
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone | Total
Number analyzed (Participants) | 302 | 153 | 455
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (9.33) | 63.7 (9.56) | 63.6 (9.40)
Age, Customized [Count of Participants; unit: Participants] — Stratification Factor 1
  Participants
    ≤ 75 Years Old | 278 | 141 | 419
    > 75 Years Old | 24 | 12 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 66 | 187
  Male | 181 | 87 | 268
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 14 | 41
  Not Hispanic or Latino | 228 | 104 | 332
  Unknown or Not Reported | 47 | 35 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 0 | 4
  Black or African American | 4 | 3 | 7
  White | 244 | 113 | 357
  Other | 2 | 2 | 4
  Not collected | 48 | 35 | 83
Participants with Prior Anti-Myeloma (MM) Therapies [Count of Participants; unit: Participants] | 302 | 153 | 455
Time from First Pathologic Diagnosis [Mean (Standard Deviation); unit: years] | 6.2 (4.02) | 6.5 (3.63) | 6.3 (3.89)
Stratification Factor 2: Disease Population [Count of Participants; unit: Participants] — Disease Population Group 1 is defined as refractory patients who have progressed on or within 60 days of both lenalidomide and bortezomib based treatments. Disease Population Group 2 is defined as relapsed and refractory patients who achieved at least a partial response (PR) and progressed within 6 months after stopping treatment with lenalidomide and/or bortezomib. Disease Population Group 3 is defined as refractory/intolerant patients who developed intolerance/toxicity after a minimum of 2 cycles of bortezomib.
  Participants
    Disease Population Group 1 | 249 | 125 | 374
    Disease Population Group 2 | 8 | 5 | 13
    Disease Population Group 3 | 45 | 23 | 68
Stratification Factor 3: Number of Prior Anti-MM Therapies [Count of Participants; unit: Participants]
  2 Prior Anti-MM Therapies | 17 | 8 | 25
  > 2 Prior Anti-MM Therapies | 285 | 145 | 430
Multiple Myeloma Stage before Study Entry [Count of Participants; unit: Participants] — The International Staging System divides myeloma into 3 stages based only on the serum beta-2 microglobulin and serum albumin levels. Stage I: Serum beta-2 microglobulin is less than 3.5 (mg/L) and the albumin level is above 3.5 (g/L); Stage II: Neither stage I or III, meaning that either: ◾ The beta-2 microglobulin level is between 3.5 and 5.5 (with any albumin level), OR ◾ The albumin is below 3.5 while the beta-2 microglobulin is less than 3.5 Stage III: Serum beta-2 microglobulin is greater than 5.5.
  Participants
    Stage I | 81 | 36 | 117
    Stage II | 115 | 56 | 171
    Stage III | 92 | 53 | 145
    Missing | 14 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) - Primary Analysis
Description: Progression-free survival was calculated as the time from randomization to disease progression as determined by the Independent Response Adjudication Committee based on the International Myeloma Working Group Uniform Response criteria (IMWG), or death on study, whichever occurred earlier. Progressive disease required 1 of the following: • Increase of ≥ 25% from nadir in: o Serum M-component (absolute increase ≥ 0.5 g/dl); o Urine M-component (absolute increase ≥ 200 mg/24 hours); o Bone marrow plasma cell percentage (absolute % ≥ 10%); • Development of new or increase in the size of existing bone lesions or soft tissue plasmacytomas; • Development of hypercalcemia (corrected serum calcium > 11.5 mg/dl) attributed solely to plasma cell proliferative disease.
Time Frame: From randomization until the data cut-off date of 07 September 2012. Maximum duration of follow-up for PFS assessments was 57 weeks.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 302 | 153
weeks | 15.7 [13.0 to 20.1] | 8.0 [7.0 to 9.0]
Statistical Analysis 1: Comparison: Pomalidomide Plus Low-Dose Dexamethasone vs High-Dose Dexamethasone; Test type: Superiority or Other; p < 0.001, Stratified Log Rank Test; Stratified by age, disease population, and prior number of anti myeloma therapy; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.35 to 0.59] — Hazard ratio is for Pomalidomide Plus Low-Dose Dexamethasone : High Dose Dexamethasone

2. Primary Outcome: Progression-free Survival (PFS) With a Later Cut-off Date
Description: Progression-free survival was calculated as the time from randomization to disease progression as determined by the Independent Response Adjudication Committee based on the International Myeloma Working Group Uniform Response criteria (IMWG), or death on study, whichever occurred earlier. Progressive disease requires 1 of the following: • Increase of ≥ 25% from nadir in: o Serum M-component (absolute increase ≥ 0.5 g/dl); o Urine M-component (absolute increase ≥ 200 mg/24 hours); o Bone marrow plasma cell percentage (absolute % ≥ 10%); • Development of new or increase in the size of existing bone lesions or soft tissue plasmacytomas; • Development of hypercalcemia (corrected serum calcium > 11.5 mg/dl) attributed solely to plasma cell proliferative disease.
Time Frame: From randomization until the data cut-off date of 01 March 2013. Maximum duration of follow-up for PFS assessments was 74 weeks.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 302 | 153
weeks | 16.0 [13.0 to 19.6] | 8.1 [7.1 to 9.4]
Statistical Analysis 1: Comparison: Pomalidomide Plus Low-Dose Dexamethasone vs High-Dose Dexamethasone; Test type: Superiority or Other; p < 0.001, Stratified log-rank test; Stratified by age, disease population, and prior number of anti myeloma therapy; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.39 to 0.61] — Hazard ratio is for Pomalidomide Plus Low-Dose Dexamethasone : High Dose Dexamethasone

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. A serious AE is any AE occurring at any dose that: • Results in death; • Is life-threatening; • Requires or prolongs existing inpatient hospitalization; • Results in persistent or significant disability/incapacity; • Is a congenital anomaly/birth defect; • Constitutes an important medical event. The Investigator assessed the relationship of each AE to study drug and graded the severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0): Grade 1 = Mild (no limitation in activity or intervention required); Grade 2 = Moderate (some limitation in activity; no/minimal medical intervention required); Grade 3 = Severe (marked limitation in activity; medical intervention required, hospitalization possible); Grade 4 = Life-threatening; Grade 5 = Death.
Time Frame: From first dose of study drug through to 30 days after the last dose as of the end of the study (29 August 2017); maximum time on treatment was 297, 269, and 239 weeks in the Pomalidomide + LD-Dex, HD-Dex, and cross-over groups respectively.
Population: Safety population (all randomized participants who received at least one dose of study drug (either pomalidomide or dexamethasone)).
Measure: Count of Participants; unit: Participants
Groups:
- High-Dose Dexamethasone: Participants received 40 mg dexamethasone (participants > 75 years of age received 20 mg dexamethasone) administered by mouth once per day on Days 1 through 4, 9 through 12, and 17 through 20 of a 28-day cycle until disease progression, or until cross-over to pomalidomide. Data are up to the time of cross-over.
- HD-Dex / Pomalidomide: Participants initially randomized to high-dose dexamethasone (HD-Dex) crossed over to receive 4 mg pomalidomide administered by mouth on Days 1-21 of each 28-day treatment cycle, with or without low-dose dexamethasone (40 mg for participants ≤ 75 years or 20 mg for participants > 75 years of age, administered orally once per day on Days 1, 8, 15, and 22 of each 28-day cycle) at the discretion of the investigator. Data include AEs that occurred after cross-over to pomalidomide.
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone | HD-Dex / Pomalidomide
Number analyzed (Participants) | 300 | 150 | 11
Participants
  Any adverse event | 298 | 149 | 11
  Grade 3-4 adverse events | 266 | 127 | 8
  AE related to pomalidomide | 251 | 0 | 11
  AE related to dexamethasone | 205 | 115 | 5
  AE related to either study drug | 271 | 115 | 11
  Grade 3-4 AE related to pomalidomide | 199 | 0 | 6
  Grade 3-4 AE related to dexamethasone | 114 | 70 | 2
  Grade 3-4 AE related to either study drug | 212 | 70 | 6
  Grade 5 adverse events | 46 | 21 | 1
  Serious adverse events (SAEs) | 195 | 80 | 4
  SAE related to pomalidomide | 89 | 0 | 1
  SAE related to dexamethasone | 73 | 36 | 0
  SAE related to either study drug | 98 | 36 | 1
  SAE leading to discontinuation of pomalidomide | 20 | 0 | 1
  SAE leading to discontinuation of dexamethasone | 20 | 14 | 1
  SAE leading to discontinuation of either study dru | 23 | 14 | 1
  AE leading to discontinuation of pomalidomide | 30 | 0 | 1
  AE leading to discontinuation of dexamethasone | 34 | 16 | 1
  AE leading to discontinuation of either study drug | 38 | 16 | 1

4. Secondary Outcome: Overall Survival - Primary Analysis
Description: Overall survival is calculated as the time from randomization to death from any cause. Overall survival was censored at the last date that the participant was known to be alive for participants who were alive at the time of analysis and for participants who were lost to follow-up before death was documented.
Time Frame: From randomization until the data cut-off date of 07 September 2012. Maximum time on follow-up for survival was 70 weeks.
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 302 | 153
weeks | NA [48.1 to NA] — Could not be estimated due to the low number of events | 34.0 [23.4 to 39.9]
Statistical Analysis 1: Comparison: Pomalidomide Plus Low-Dose Dexamethasone vs High-Dose Dexamethasone; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.37 to 0.74] — Hazard ratio is for Pomalidomide Plus Low-Dose Dexamethasone : High Dose Dexamethasone

5. Secondary Outcome: Overall Survival With a Later Cut-off Date
Description: as for outcome 4
Time Frame: From randomization until the data cut-off date of 01 March 2013. Maximum time on follow-up for survival was 93 weeks.
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 302 | 153
weeks | 54.0 [45.3 to 66.4] | 34.9 [29.9 to 39.1]
Statistical Analysis 1: Comparison: Pomalidomide Plus Low-Dose Dexamethasone vs High-Dose Dexamethasone; Test type: Superiority or Other; p = 0.009, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.54 to 0.92] — Hazard ratio is for Pomalidomide Plus Low-Dose Dexamethasone : High Dose Dexamethasone

6. Secondary Outcome: Overall Survival Based on the Final Dataset
Description: as for outcome 4
Time Frame: From randomization until the data cut-off date of 29 August 2017. Maximum time on follow-up for survival was 324 weeks.
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 302 | 153
weeks | 56.1 [47.7 to 67.4] | 35.3 [29.9 to 39.9]
Statistical Analysis 1: Comparison: Pomalidomide Plus Low-Dose Dexamethasone vs High-Dose Dexamethasone; Test type: Superiority; p = 0.005, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.60 to 0.91] — Hazard ratio is for Pomalidomide Plus Low-Dose Dexamethasone : High Dose Dexamethasone

7. Secondary Outcome: Percentage of Participants With an Objective Response According to International Myeloma Working Group (IMWG) Uniform Response Criteria
Description: Objective response is defined as a best overall response of stringent complete response (SCR), complete response (CR), very good partial response (VGPR) or partial response (PR) based on the Independent Response Adjudication Committee: SCR: CR and normal free light chain (FLC) ratio and no clonal cells in bone marrow; CR: Negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein and urine M-protein level < 100 mg/24 hours; PR: ≥ 50% reduction of serum M-Protein and reduction in urinary M-protein by ≥ 90% or to < 200 mg/24 hours. In addition to the above, if present at baseline a ≥ 50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: From randomization until the data cut-off date of 01 March 2013. Maximum time on follow-up was 93 weeks.
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 302 | 153
percentage of participants | 23.5 | 3.9
Statistical Analysis 1: Comparison: Pomalidomide Plus Low-Dose Dexamethasone vs High-Dose Dexamethasone; Test type: Superiority or Other; p < 0.001, Fisher Exact; Odds Ratio (OR) = 7.53, 95% CI 2-sided [3.19 to 17.77] — Odds ratio is for pomalidomide plus low-dose dexamethasone : high dose dexamethasone

8. Secondary Outcome: Percentage of Participants With Objective Response According to European Group for Blood and Marrow Transplantation (EBMT) Criteria
Description: Objective response defined as a best overall response of complete response (CR) or partial response (PR) based on the Independent Response Adjudication Committee: CR requires all of the following: - Absence of original monoclonal paraprotein in serum and urine by immunofixation maintained at least 42 days. - <5% plasma cell in bone marrow aspirate and on bone marrow biopsy, if performed. - No increase in size or number of lytic bone lesions. - Disappearance of soft tissue plasmacytomas. PR requires all of the following: - ≥ 50% reduction in level of serum monoclonal paraprotein, maintained at least 42 days. - Reduction in 24-hour urinary light chain extraction by ≥ 90% or to < 200 mg, maintained at least 42 days. - For patients with non-secretory myeloma, ≥ 50% reduction in plasma cells in bone marrow aspirate and on biopsy, if performed, for at least 42 days. - ≥ 50% reduction in the size of soft tissue plasmacytomas. - No increase in size or number of lytic bone lesions.
Time Frame: From randomization until the data cut-off date of 01 March 2013. Maximum time on follow-up was 93 weeks.
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 302 | 153
percentage of participants | 22.2 | 3.3
Statistical Analysis 1: Comparison: Pomalidomide Plus Low-Dose Dexamethasone vs High-Dose Dexamethasone; Test type: Superiority or Other; p < 0.001, Fisher Exact; Odds Ratio (OR) = 8.44, 95% CI 2-sided [3.32 to 21.42] — Odds ratio is for Pomalidomide Plus Low-Dose Dexamethasone : High Dose Dexamethasone

9. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) is calculated as the time from randomization to the first documented progression confirmed by a blinded, independent Response Adjudication Committee and based on the International Myeloma Working Group Uniform Response criteria (IMWG). Progressive disease requires 1 of the following: • Increase of ≥ 25% from nadir in: o Serum M-component (absolute increase ≥ 0.5 g/dl); o Urine M-component (absolute increase ≥ 200 mg/24 hours); o Bone marrow plasma cell percentage (absolute % ≥ 10%); • Development of new or increase in the size of existing bone lesions or soft tissue plasmacytomas; • Development of hypercalcemia (corrected serum calcium > 11.5 mg/dl) attributed solely to plasma cell proliferative disease.
Time Frame: From randomization until the data cut-off date of 01 March 2013. Maximum time on follow-up was 93 weeks.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 302 | 153
weeks | 20.0 [16.1 to 24.0] | 9.0 [8.0 to 10.9]
Statistical Analysis 1: Comparison: Pomalidomide Plus Low-Dose Dexamethasone vs High-Dose Dexamethasone; Test type: Superiority or Other; p < 0.001, Stratified Log Rank Test; Stratified by age, diseases population, and prior number of anti myeloma therapy; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.36 to 0.59] — Hazard ratio is for Pomalidomide Plus Low-Dose Dexamethasone : High Dose Dexamethasone

10. Secondary Outcome: Time to Response
Description: Time to response is calculated as the time from randomization to the initial documented response (partial response or better) based on IMWG criteria. SCR: CR and normal free light chain (FLC) ratio and no clonal cells in bone marrow; CR: Negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein and urine M-protein level < 100 mg/24 hours; PR: ≥ 50% reduction of serum M-Protein and reduction in urinary M-protein by ≥ 90% or to < 200 mg/24 hours. If present at baseline a ≥ 50% reduction in size of soft tissue plasmacytomas is also required.
Time Frame: From randomization until the data cut-off date of 01 March 2013. Maximum time on follow-up was 93 weeks.
Population: Intent-to-treat responder population
Measure: Median (Full Range); unit: weeks
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 71 | 6
weeks | 8.1 [4.0 to 48.0] | 10.5 [4.1 to 42.1]

11. Secondary Outcome: Duration of Response
Description: Duration of response (calculated for responders only) is defined as time from the initial documented response (partial response or better) to confirmed disease progression, based on IMWG criteria assessed by the Independent Response Adjudication Committee.
Time Frame: From randomization until the data cut-off date of 01 March 2013. Maximum time on follow-up was 93 weeks.
Population: Intent-to-treat responder population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 71 | 6
weeks | 35.1 [28.4 to 52.9] | 28.1 [20.1 to 37.1]

12. Secondary Outcome: Time to the First Hemoglobin Improvement
Description: Time to increased hemoglobin, defined as the time from randomization to at least one category improvement from Baseline in common terminology criteria for adverse events (CTCAE) grade for hemoglobin level. Hemoglobin categories are: 1) Normal; 2) CTCAE Grade 1: < lower limit of normal (LLN) to 10.0 g/dL; 3) CTCAE Grade 2: < 10.0 to <8.0 g/dL. Participants with CTCAE Grade 3 anemia or worse at Baseline were excluded from the study.
Time Frame: From randomization until the data cut-off date of 01 March 2013. Maximum time on follow-up was 93 weeks.
Population: Intent-to-treat population with improvement in hemoglobin during the study
Measure: Median (Full Range); unit: weeks
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 144 | 50
weeks | 3.4 [1.1 to 49.3] | 1.3 [0.9 to 24.3]

13. Secondary Outcome: Time to Improvement in Bone Pain
Description: Time to improvement in bone pain is defined as the time from randomization to at least one category improvement from Baseline in bone pain category. Bone pain was categorized (from best to worst) according to answers to the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire for patients with Multiple Myeloma Module (QLQ-MY20), Question 1, "Have you had bone aches or pain?": 1) Not at all, 2) A little, 3) Quite a bit, or 4) Very much.
Time Frame: From randomization until the data cut-off date of 01 March 2013. Maximum time on follow-up was 93 weeks.
Population: Intent-to-treat population with improvement in bone pain
Measure: Median (Full Range); unit: weeks
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 101 | 37
weeks | 5.7 [3.7 to 88.6] | 4.1 [3.7 to 27.3]

14. Secondary Outcome: Time to Improvement in Renal Function
Description: Time to improvement in renal function is defined as the time from randomization to at least one category improvement from Baseline in renal function. Renal Function was categorized as (from best to worst): - Normal: creatinine clearance ≥80 mL/min; - Grade 1: creatinine clearance ≥60 to <80 mL/min; - Grade 2 : creatinine clearance ≥45 to < 60 mL/min. Participants with creatinine clearance < 45 mL/min at baseline were excluded from the study.
Time Frame: From randomization until the data cut-off date of 01 March 2013. Maximum time on follow-up was 93 weeks.
Population: Intent-to-treat population with improvement in renal function
Measure: Median (Full Range); unit: weeks
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 94 | 45
weeks | 4.6 [3.3 to 45.6] | 4.1 [3.3 to 28.1]

15. Secondary Outcome: Time to Improvement in Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: Time to improvement in ECOG performance status defined as the time from randomization until at least a one category improvement from Baseline in ECOG performance status score. The categories of the ECOG Performance Status Scale are as follows: -0: Fully active, able to carry on all pre-disease performance without restriction; -1: Restricted in physically strenuous activity but ambulatory and able to carry our work of a light or sedentary nature, e.g., light housework, office work; -2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours. Patients with a score of 3, 4 or 5 were excluded from participating in the study.
Time Frame: From randomization until the data cut-off date of 01 March 2013. Maximum time on follow-up was 93 weeks.
Population: Intent-to-treat population with improvement in ECOG performance status during the study
Measure: Median (Full Range); unit: weeks
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 61 | 18
weeks | 8.1 [4.1 to 44.1] | 4.3 [4.1 to 33.7]

16. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Global Health Status Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Global Health Status/QOL scale is scored between 0 and 100, with a high score indicating better Global Health Status/QOL. Negative change from Baseline values indicate deterioration in QOL or functioning and positive values indicate improvement.
Time Frame: Day 1 of Cycle 1 (Baseline), and Day 1 of Cycles 2, 3, 4, 5 and 6
Population: The Patient Reported Outcomes (PRO) study population includes any intent-to-treat study participants with 1 active treatment and 1 PRO measurement item completed. Only participants with available data at Baseline and each time point are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 289 | 144
units on a scale
  Cycle 2, Day 1: number analyzed (Participants) | 209 | 91
  Cycle 2, Day 1 | 0.52 (23.01) | -3.75 (24.10)
  Cycle 3, Day 1: number analyzed (Participants) | 175 | 53
  Cycle 3, Day 1 | 2.67 (24.97) | -2.36 (21.08)
  Cycle 4, Day 1: number analyzed (Participants) | 157 | 33
  Cycle 4, Day 1 | 0.80 (24.62) | -3.03 (22.42)
  Cycle 5 Day 1: number analyzed (Participants) | 130 | 27
  Cycle 5 Day 1 | 0.51 (26.81) | 0.00 (27.44)
  Cycle 6, Day 1: number analyzed (Participants) | 116 | 18
  Cycle 6, Day 1 | -2.51 (25.57) | -0.93 (17.59)

17. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Physical Functioning Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Physical Functioning Scale is scored between 0 and 100, with a high score indicating better functioning/support. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: Day 1 of Cycle 1 (Baseline), and Day 1 of Cycles 2, 3, 4, 5 and 6
Population: PRO population with available data at Baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 289 | 144
units on a scale
  Cycle 2, Day 1: number analyzed (Participants) | 210 | 91
  Cycle 2, Day 1 | -2.32 (18.25) | -3.96 (18.35)
  Cycle 3, Day 1: number analyzed (Participants) | 177 | 53
  Cycle 3, Day 1 | -0.56 (19.86) | -9.69 (16.67)
  Cycle 4, Day 1: number analyzed (Participants) | 159 | 33
  Cycle 4, Day 1 | 0.17 (20.25) | -8.08 (13.31)
  Cycle 5 Day 1: number analyzed (Participants) | 132 | 27
  Cycle 5 Day 1 | 0.91 (19.92) | -5.43 (19.31)
  Cycle 6, Day 1: number analyzed (Participants) | 118 | 18
  Cycle 6, Day 1 | 0.54 (21.30) | -4.81 (14.24)

18. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Emotional Functioning Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Emotional Functioning Scale is scored between 0 and 100, with a high score indicating better functioning/support. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: Day 1 of Cycle 1 (Baseline), and Day 1 of Cycles 2, 3, 4, 5 and 6
Population: PRO population with available data at Baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 289 | 144
units on a scale
  Cycle 2, Day 1: number analyzed (Participants) | 210 | 91
  Cycle 2, Day 1 | 1.22 (21.44) | -2.87 (21.57)
  Cycle 3, Day 1: number analyzed (Participants) | 176 | 53
  Cycle 3, Day 1 | 2.40 (20.36) | -5.66 (25.36)
  Cycle 4, Day 1: number analyzed (Participants) | 158 | 33
  Cycle 4, Day 1 | 2.44 (21.05) | -6.31 (23.48)
  Cycle 5 Day 1: number analyzed (Participants) | 131 | 27
  Cycle 5 Day 1 | 1.91 (21.97) | -8.64 (23.17)
  Cycle 6, Day 1: number analyzed (Participants) | 117 | 18
  Cycle 6, Day 1 | 0.19 (22.30) | -4.17 (13.18)

19. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Fatigue Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Fatigue Scale is scored between 0 and 100, with a high score indicating a higher level of symptoms. Negative change from Baseline values indicate reduction in fatigue (i.e. improvement in symptom) and positive values indicate increases in fatigue (i.e. worsening of symptom).
Time Frame: Day 1 of Cycle 1 (Baseline), and Day 1 of Cycles 2, 3, 4, 5 and 6
Population: PRO population with available data at Baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 289 | 144
units on a scale
  Cycle 2, Day 1: number analyzed (Participants) | 210 | 91
  Cycle 2, Day 1 | 2.43 (27.39) | 4.03 (25.37)
  Cycle 3, Day 1: number analyzed (Participants) | 177 | 53
  Cycle 3, Day 1 | 3.26 (27.66) | 7.76 (23.73)
  Cycle 4, Day 1: number analyzed (Participants) | 159 | 33
  Cycle 4, Day 1 | 1.71 (26.21) | 9.43 (28.88)
  Cycle 5 Day 1: number analyzed (Participants) | 132 | 27
  Cycle 5 Day 1 | 0.21 (28.41) | 9.47 (23.00)
  Cycle 6, Day 1: number analyzed (Participants) | 118 | 18
  Cycle 6, Day 1 | 0.99 (31.13) | 10.49 (16.38)

20. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Pain Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Pain Scale is scored between 0 and 100, with a high score indicating a higher level of symptoms. Negative change from Baseline values indicate reductions in pain (i.e. improvement in symptom) and positive values indicate increases in pain (i.e. worsening of symptom).
Time Frame: Day 1 of Cycle 1 (Baseline), and Day 1 of Cycles 2, 3, 4, 5 and 6
Population: PRO population with available data at Baseline and each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 289 | 144
units on a scale
  Cycle 2, Day 1: number analyzed (Participants) | 210 | 92
  Cycle 2, Day 1 | -2.70 (25.74) | 0.36 (25.32)
  Cycle 3, Day 1: number analyzed (Participants) | 177 | 53
  Cycle 3, Day 1 | -3.58 (29.62) | 2.83 (25.47)
  Cycle 4, Day 1: number analyzed (Participants) | 159 | 33
  Cycle 4, Day 1 | -2.41 (30.52) | 3.03 (25.84)
  Cycle 5 Day 1: number analyzed (Participants) | 132 | 27
  Cycle 5 Day 1 | -1.64 (28.00) | 2.47 (31.59)
  Cycle 6, Day 1: number analyzed (Participants) | 118 | 18
  Cycle 6, Day 1 | -2.40 (30.99) | 10.19 (23.67)

21. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer QoL Questionnaire for Patients With Multiple Myeloma (EORTC QLQ-MY20) Disease Symptoms
Description: The European Organization for Research and Treatment of Cancer QoL Questionnaire for Patients with Multiple Myeloma (EORTC QLQ-MY20) is a 20-question tool used in clinical research to assess health-related quality of life in multiple myeloma patients. The QLQ-MY20 includes four domains (Disease Symptoms, Side-Effects of Treatment, Body Image and Future Perspective). The EORTC QLQ-MY20 Disease Symptoms Scale is scored between 0 and 100, with a high score reflecting a higher level of symptoms. Negative change from Baseline values indicate reduction (i.e. improvement) in symptoms and positive values indicate increase (i.e. worsening) of symptoms.
Time Frame: Day 1 of Cycle 1 (Baseline), and Day 1 of Cycles 2, 3, 4, 5 and 6
Population: PRO population with available data at Baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 289 | 144
units on a scale
  Cycle 2, Day 1: number analyzed (Participants) | 218 | 99
  Cycle 2, Day 1 | -0.50 (16.51) | -1.07 (17.78)
  Cycle 3, Day 1: number analyzed (Participants) | 180 | 56
  Cycle 3, Day 1 | -1.36 (19.51) | 0.97 (19.93)
  Cycle 4, Day 1: number analyzed (Participants) | 161 | 37
  Cycle 4, Day 1 | -1.15 (19.54) | 1.35 (16.94)
  Cycle 5 Day 1: number analyzed (Participants) | 135 | 30
  Cycle 5 Day 1 | -0.53 (17.39) | 1.48 (17.56)
  Cycle 6, Day 1: number analyzed (Participants) | 115 | 21
  Cycle 6, Day 1 | 0.60 (19.64) | 2.12 (13.43)

22. Secondary Outcome: Change From Baseline in the EORTC QLQ-MY20 Side Effects Domain
Description: The European Organization for Research and Treatment of Cancer QoL Questionnaire for Patients with Multiple Myeloma (EORTC QLQ-MY20) is a 20-question tool used in clinical research to assess health-related quality of life in multiple myeloma patients. The QLQ-MY20 includes four domains (Disease Symptoms, Side-Effects of Treatment, Body Image and Future Perspective). The EORTC QLQ-MY20 Side Effects Scale is scored between 0 and 100, with a high score reflecting a higher level of symptoms. Negative change from Baseline values indicate reduction in side effects (i.e.improvement in symptom) and positive values indicate increase in side effects (i.e. worsening of symptom).
Time Frame: Day 1 of Cycle 1 (Baseline), and Day 1 of Cycles 2, 3, 4, 5 and 6
Population: PRO population with available data at Baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 289 | 144
units on a scale
  Cycle 2, Day 1: number analyzed (Participants) | 218 | 99
  Cycle 2, Day 1 | 2.71 (13.90) | 2.61 (13.34)
  Cycle 3, Day 1: number analyzed (Participants) | 180 | 55
  Cycle 3, Day 1 | 3.26 (13.72) | 5.35 (12.27)
  Cycle 4, Day 1: number analyzed (Participants) | 161 | 37
  Cycle 4, Day 1 | 3.73 (14.47) | 7.46 (11.61)
  Cycle 5 Day 1: number analyzed (Participants) | 135 | 30
  Cycle 5 Day 1 | 4.74 (14.45) | 6.89 (10.32)
  Cycle 6, Day 1: number analyzed (Participants) | 115 | 21
  Cycle 6, Day 1 | 4.55 (15.76) | 7.30 (9.35)

23. Secondary Outcome: Change From Baseline in the European Quality of Life-5 Dimensions (EQ-5D) Utility Index Score
Description: EQ-5D is a self-administered questionnaire that assesses health-related quality of life (QOL). The EQ-5D descriptive health profile comprises five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension has 3 levels of response: No problem (1), some problems (2), and extreme problems (3). A unique EQ-5D health state is defined by combining one level from each of the five dimensions into a single utility index score. EQ-5D index values range from -0.59 to 1.00 where an EQ-5D score of 1.00 equals "perfect health", a score of 0 equals "death" and a score of -0.59 equals worst imaginable health state. A positive change from Baseline score indicates improvement in health status. A negative change from Baseline score indicates worsening in health status. Negative scores represent the possible though unlikely situation that a patient's QOL is worse than death, i.e. they would rather be dead than living with that QOL
Time Frame: Day 1 of Cycle 1 (Baseline), and Day 1 of Cycles 2, 3, 4, 5 and 6
Population: PRO population with available data at Baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 289 | 144
units on a scale
  Cycle 2, Day 1: number analyzed (Participants) | 198 | 89
  Cycle 2, Day 1 | -0.03 (0.28) | -0.02 (0.23)
  Cycle 3, Day 1: number analyzed (Participants) | 167 | 52
  Cycle 3, Day 1 | 0.01 (0.29) | -0.06 (0.27)
  Cycle 4, Day 1: number analyzed (Participants) | 146 | 33
  Cycle 4, Day 1 | 0.04 (0.31) | -0.07 (0.29)
  Cycle 5, Day 1: number analyzed (Participants) | 125 | 25
  Cycle 5, Day 1 | 0.01 (0.32) | -0.04 (0.26)
  Cycle 6, Day 1: number analyzed (Participants) | 108 | 18
  Cycle 6, Day 1 | 0.03 (0.31) | -0.12 (0.19)

24. Secondary Outcome: Time to First Worsening of Quality of Life (QOL) Domains
Description: Time to worsening in quality of life domains was calculated as the time from Baseline to the first worsened minimally important difference (MID), defined as the smallest change in a QOL score considered important to patients that would lead the patient or clinician to consider a change in therapy. MID thresholds were calculated in Standard Error of Measurement (SEM) units using the Baseline QOL data. Based on the MID, participants were classified as worsened according to the following: For the EORTC QLQ-C30 global health status and functional scales and the EQ-5D health utility score, participants were classified as worsened if their change from Baseline score was less than -1 SEM. For the EORTC QLQ-C30 symptom scores (fatigue and pain) and EORTC QLQ-MY20 disease symptoms and side effects scales, participants were classified as worsened if their change from Baseline score was greater than 1 SEM. See previous outcome measures for definitions of each scale.
Time Frame: Assessed on Day 1 of the first 6 treatment cycles.
Population: PRO population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone
Number analyzed (Participants) | 289 | 144
days
  Global Health Status | 71 [60 to 92] | 57 [36 to 91]
  Physical Functioning | 128 [92 to 225] | 67 [57 to 106]
  Emotional Functioning | 146 [120 to 259] | 85 [57 to 124]
  Fatigue | 58 [57 to 85] | 57 [46 to 67]
  Pain | 92 [86 to 147] | 85 [62 to 337]
  Disease Symptoms | 127 [92 to 155] | 106 [67 to 141]
  Side Effects of Treatment | 90 [78 to 123] | 85 [58 to 113]
  Health Utility | 225 [123 to 338] | 162 [85 to NA] — Could not be calculated due to a low number of events

ADVERSE EVENTS:
Time Frame: From first dose of study drug through to 30 days after the last dose as of the end of the study (29 August 2017); maximum time on treatment was 297, 269, and 239 weeks in the Pomalidomide + LD-Dex, HD-Dex, and cross-over groups respectively.
Arm/Group | Pomalidomide Plus Low-Dose Dexamethasone | High-Dose Dexamethasone | HD-Dex / Pomalidomide
All-Cause Mortality (participants affected / at risk) | 252/300 | 124/150 | 8/11
Serious Adverse Events (participants affected / at risk) | 195/300 | 80/150 | 4/11
Other Adverse Events (participants affected / at risk) | 291/300 | 143/150 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide Plus Low-Dose Dexamethasone (N=300) | High-Dose Dexamethasone (N=150) | HD-Dex / Pomalidomide (N=11)
Anaemia (Blood and lymphatic system disorders) | 10 | 7 | 0
Blood disorder (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 19 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 10 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 4 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac amyloidosis (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 1
Cardiac failure (Cardiac disorders) | 4 | 2 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Necrotising colitis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Papilla of Vater stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 2 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 0
General physical health deterioration (General disorders) | 26 | 12 | 0
Hyperthermia (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 2 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 4 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 2 | 0 | 0
Performance status decreased (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 26 | 7 | 0
Sudden death (General disorders) | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic mass (Hepatobiliary disorders) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Aspergillus infection (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 2 | 1 | 0
Bacterial diarrhoea (Infections and infestations) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 8 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 2 | 0 | 0
Device related infection (Infections and infestations) | 3 | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Enterobacter infection (Infections and infestations) | 1 | 0 | 0
Enterobacter sepsis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 3 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 1 | 0
Infection (Infections and infestations) | 3 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0
Listeria sepsis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 6 | 4 | 1
Lung infection (Infections and infestations) | 5 | 1 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0
Meningitis cryptococcal (Infections and infestations) | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 3 | 0 | 0
Ophthalmic herpes simplex (Infections and infestations) | 0 | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0
Pneumococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 | 1 | 0
Pneumonia (Infections and infestations) | 57 | 14 | 2
Pneumonia bacterial (Infections and infestations) | 2 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 1 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 4 | 0 | 1
Salmonella sepsis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 7 | 3 | 0
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0
Septic arthritis streptococcal (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 4 | 6 | 0
Sialoadenitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Spinal cord infection (Infections and infestations) | 1 | 0 | 0
Streptococcal infection (Infections and infestations) | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Subdural empyema (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 5 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 5 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 2 | 0
Blood immunoglobulin M increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 13 | 5 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 1 | 0
Coma (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Dyspraxia (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 2 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Vertigo CNS origin (Nervous system disorders) | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0
Bradyphrenia (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 3 | 3 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 11 | 7 | 1
Crush syndrome (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 8 | 1 | 0
Renal impairment (Renal and urinary disorders) | 4 | 2 | 0
Urinary retention (Renal and urinary disorders) | 3 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Axillary vein thrombosis (Vascular disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide Plus Low-Dose Dexamethasone (N=300) | High-Dose Dexamethasone (N=150) | HD-Dex / Pomalidomide (N=11)
Anaemia (Blood and lymphatic system disorders) | 159 | 77 | 4
Leukopenia (Blood and lymphatic system disorders) | 40 | 8 | 0
Lymphopenia (Blood and lymphatic system disorders) | 13 | 8 | 0
Neutropenia (Blood and lymphatic system disorders) | 155 | 30 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 87 | 42 | 1
Palpitations (Cardiac disorders) | 7 | 4 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 2 | 1 | 1
Cataract (Eye disorders) | 8 | 4 | 1
Macular pigmentation (Eye disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 8 | 3 | 1
Constipation (Gastrointestinal disorders) | 72 | 22 | 1
Diarrhoea (Gastrointestinal disorders) | 73 | 26 | 3
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 3 | 2 | 1
Nausea (Gastrointestinal disorders) | 57 | 16 | 3
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 25 | 6 | 1
Asthenia (General disorders) | 53 | 25 | 1
Chest pain (General disorders) | 11 | 4 | 1
Chills (General disorders) | 18 | 2 | 0
Fatigue (General disorders) | 103 | 40 | 3
General physical health deterioration (General disorders) | 17 | 5 | 0
Influenza like illness (General disorders) | 3 | 1 | 2
Malaise (General disorders) | 10 | 1 | 1
Oedema (General disorders) | 9 | 7 | 1
Oedema peripheral (General disorders) | 51 | 15 | 3
Pyrexia (General disorders) | 74 | 31 | 3
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 34 | 7 | 1
Cellulitis (Infections and infestations) | 6 | 2 | 1
Herpes zoster (Infections and infestations) | 6 | 1 | 1
Nasopharyngitis (Infections and infestations) | 30 | 1 | 1
Pneumonia (Infections and infestations) | 19 | 5 | 0
Respiratory tract infection (Infections and infestations) | 15 | 5 | 0
Sinusitis (Infections and infestations) | 10 | 4 | 1
Tooth abscess (Infections and infestations) | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 47 | 10 | 2
Urinary tract infection (Infections and infestations) | 18 | 6 | 2
Wound infection (Infections and infestations) | 0 | 0 | 1
Chillblains (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 5 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 10 | 4 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 7 | 2 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 18 | 6 | 2
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 19 | 1 | 1
Weight decreased (Investigations) | 15 | 5 | 2
White blood cell count decreased (Investigations) | 10 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 40 | 10 | 3
Dehydration (Metabolism and nutrition disorders) | 14 | 8 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 11 | 11 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 18 | 10 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 14 | 9 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 31 | 12 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 7 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 59 | 23 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 54 | 20 | 2
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 47 | 11 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 | 18 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12 | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 18 | 5 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 4 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 4 | 11 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 9 | 0
Amnesia (Nervous system disorders) | 2 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 40 | 13 | 0
Headache (Nervous system disorders) | 28 | 9 | 1
Lethargy (Nervous system disorders) | 9 | 4 | 1
Neuropathy peripheral (Nervous system disorders) | 9 | 1 | 1
Paraesthesia (Nervous system disorders) | 12 | 6 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 26 | 4 | 2
Tremor (Nervous system disorders) | 19 | 2 | 0
Agitation (Psychiatric disorders) | 17 | 7 | 0
Anxiety (Psychiatric disorders) | 15 | 9 | 0
Confusional state (Psychiatric disorders) | 10 | 7 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 36 | 32 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 3 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 64 | 15 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 60 | 21 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 18 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 26 | 13 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 8 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 18 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 25 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 4 | 1
Haematoma (Vascular disorders) | 9 | 2 | 1
Hot flush (Vascular disorders) | 2 | 2 | 1
Hypotension (Vascular disorders) | 13 | 4 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution may publish the results of its findings if a multicenter publication is not forthcoming within 18 months after study completion. Institution shall provide Celgene with a copy of the papers prior to submission; Celgene shall complete its review within 60 days after receipt. Upon Celgene's request, proposed publication or presentation will be delayed up to 60 additional days to enable Celgene to secure adequate intellectual property protection of patentable material.